CLINICAL TRIAL: NCT04855760
Title: A Phase 3, Multicenter, Open-Label Study to Assess the Long-Term Safety of REL-1017 as a Treatment of Major Depressive Disorder
Brief Title: Safety of REL-1017 for Major Depressive Disorder
Acronym: RELIANCE-OLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REL-1017-310
Expanded Access: NCT06009003 (Temporarily not available)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder
Keywords: REL-1017
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REL-1017 (Experimental): Roll-over participants received 25 mg REL-1017 (one 25 mg REL-1017 tablet), orally, per day, either as a monotherapy or in addition to their ongoing antidepressant (ADT), rolling over from the monotherapy study REL-1017-303 or the adjunctive therapy studies REL-1017-301 and REL-1017-302, respectively.
  De Novo participants received a 75 mg REL-1017 loading dose (three 25 mg REL-1017 tablets) on Day-1 of the 365-day treatment period. From Day-2 to Day-365, participants received 25 mg REL-1017 either as monotherapy or as adjunctive therapy.
  Interventions: Drug: REL-1017

INTERVENTIONS:
Drug: REL-1017 — REL-1017 tablet
  Other Names: Esmethadone HCl

SUMMARY:
This was a 1-year, multicenter, open-label, long-term study to assess the safety of REL-1017 once daily (QD) as monotherapy or as adjunctive treatment of Major Depressive Disorder. Adjunctive study participants continued to take their current antidepressant therapy in addition to the study drug for the duration of the treatment period.

DETAILED DESCRIPTION:
This was a multicenter, open-label, long-term study of REL-1017 to evaluate the long-term safety and long-term durability of response in patients with MDD. Patients who completed previous randomized, double-blind Phase 3 trials (NCT04688164, NCT04855747, NCT05081167) of REL-1017 as adjunctive therapy or monotherapy for MDD were asked to continue treatment with REL-1017 25 mg daily for up to 1 year. De novo patients who satisfied inclusion/exclusion criteria also were enrolled and received a 75 mg loading dose of REL-1017 on Day 1 followed by a maintenance dose of 25 mg REL-1017 daily for the remainder of the study (Days 2-365). When REL-1017 was administered as adjunctive treatment, patients continued to use a stable dosage of their concomitant antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 65 years, inclusive.
* Diagnosed with Major Depressive Disorder (MDD) based on Structured Clinical Interview for DSM-5 (SCID-5) for MDD.
* Current major depressive episode.

Exclusion Criteria:

* Any current and primary psychiatric disorder other than Major Depressive Disorder.
* History of bipolar I and II disorder, psychosis, and/or mania.
* Acute or chronic condition that, in the Investigator's opinion, would limit the subject's ability to complete or participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pappagallo, MD, Study Director — Relmada Therapeutics
Locations (7):
- United States (7):
  - Relmada Site, Miami, Florida
  - Relmada Site, Orlando, Florida
  - Relmada Site, Palm Bay, Florida
  - Relmada Site, Chicago, Illinois
  - Relmada Site, Boston, Massachusetts
  - Relmada Site, Watertown, Massachusetts
  - Relmada Site, Staten Island, New York

REFERENCES:
- [Derived] Fava M, Pani L, De Martin S, Cutler AJ, Gorodetzky CW, Vocci FJ, Sapienza FL, Kosten TR, Kroger C, Champasa P, Guidetti C, Comai S, Mattarei A, Folli F, Bushnell D, Traversa S, Inturrisi CE, Manfredi PL, Pappagallo M. Long-Term Safety and Efficacy of Esmethadone in Patients With Major Depressive Disorder: Findings From a 12-Month Open-Label Study. J Clin Psychiatry. 2025 Feb 17;86(1):24m15438. doi: 10.4088/JCP.24m15438. PMID 39999772

RESULTS

PARTICIPANT FLOW:
Groups:
- REL-1017: Roll-over participants received 25 mg REL-1017 (one 25 mg REL-1017 tablet), orally, per day, either as a monotherapy or in addition to their ongoing antidepressant (ADT), rolling over from the monotherapy study REL-1017-303 or the adjunctive therapy studies REL-1017-301 and REL-1017-302, respectively.
  De Novo participants received a 75 mg REL-1017 loading dose (three 25 mg REL-1017 tablets) on Day-1 of the 365-day treatment period. From Day-2 to Day-365, participants received 25 mg REL-1017 either as monotherapy or as adjunctive therapy.
  REL-1017: REL-1017 tablet
Period: Overall Study
Arm/Group | REL-1017
Started | 627
Dosed | 624
Completed | 182
Not Completed | 445
Not completed — Adverse Event | 21
Not completed — Withdrawal by Subject | 116
Not completed — Lack of Efficacy | 21
Not completed — Lost to Follow-up | 49
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 5
Not completed — Pregnancy | 1
Not completed — Non-Compliance with Study Drug | 11
Not completed — Non-Compliance with Study Schedule | 4
Not completed — Study Completed by Sponsor | 202
Not completed — Other | 13

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug.
Groups:
- REL-1017: Total participants in Open Label Study, including:
  Roll-over participants, rolling over from the monotherapy study REL-1017-303 or the adjunctive therapy studies REL-1017-301 and REL-1017-302, respectively.
  De Novo participants receiving REL1017 as either monotherapy or as adjunctive therapy.
  REL-1017: REL-1017 tablet
Arm/Group | REL-1017
Number analyzed (Participants) | 624
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 433
  Male | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 162
  Not Hispanic or Latino | 442
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 95
  White | 474
  More than one race | 16
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of REL-1017 as Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: Subjects with at least one Treatment Emergent Adverse Events (TEAEs)
Time Frame: 52 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- REL-1017: Total participants in Open Label Study
  REL-1017: REL-1017 tablet
Arm/Group | REL-1017
Number analyzed (Participants) | 624
participants | 350

2. Secondary Outcome: Change in the QT Interval With Fridericia's Correction (QTcF) Interval From Baseline to Month 3
Description: Cardiac Safety of REL-1017 as measured by the Change in the QT interval with Fridericia's correction (QTcF) Interval From Baseline to Month 3.
  A negative change from baseline indicates shortening of the QTcF.
Time Frame: 3 Month
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug and were assessed for the secondary safety endpoint at both Baseline and Month 3.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | REL-1017
Number analyzed (Participants) | 534
ms | 4.11 (14.54)

3. Secondary Outcome: Change in the QT Interval With Fridericia's Correction (QTcF) Interval From Baseline to Month 6
Description: Cardiac Safety of REL-1017 as measured by the Change in the QT interval with Fridericia's correction (QTcF) Interval From Baseline to Month 6.
  A negative change from baseline indicates shortening of the QTcF.
Time Frame: 6 Month
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug and were assessed for the secondary safety endpoint at both Baseline and Month 6.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | REL-1017
Number analyzed (Participants) | 435
ms | 2.70 (15.26)

4. Secondary Outcome: Change in the QT Interval With Fridericia's Correction (QTcF) Interval From Baseline to Month 12
Description: Cardiac Safety of REL-1017 as measured by the Change in the QT interval with Fridericia's correction (QTcF) Interval From Baseline to Month 12.
  A negative change from baseline indicates shortening of the QTcF.
Time Frame: 12 Month
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug and were assessed for the secondary safety endpoint at both Baseline and Month 12.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | REL-1017
Number analyzed (Participants) | 198
ms | 2.59 (13.77)

5. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Month 3
Description: Cardiac Safety of REL-1017 as measured by the Diastolic Blood Pressure (Supine/Semi-Supine) From Baseline to Month 3.
  A negative change from baseline indicates a reduction in Diastolic Blood Pressure.
Time Frame: 3 Month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | REL-1017
Number analyzed (Participants) | 505
mmHg | 0.5 (7.3)

6. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Month 12
Description: Cardiac Safety of REL-1017 as measured by the Diastolic Blood Pressure (Supine/Semi-Supine) From Baseline to Month 12.
  A negative change from baseline indicates a reduction in Diastolic Blood Pressure.
Time Frame: 12 Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | REL-1017
Number analyzed (Participants) | 186
mmHg | -0.2 (8.4)

7. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Month 3
Description: Cardiac Safety of REL-1017 as measured by the Systolic Blood Pressure (Supine/Semi-Supine) From Baseline to Month 3.
  A negative change from baseline indicates a reduction in Systolic Blood Pressure.
Time Frame: 3 Month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | REL-1017
Number analyzed (Participants) | 505
mmHg | 0.4 (9.9)

8. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Month 12
Description: Cardiac Safety of REL-1017 as measured by the Systolic Blood Pressure (Supine/Semi-Supine) From Baseline to Month 12.
  A negative change from baseline indicates a reduction in Systolic Blood Pressure.
Time Frame: 12 Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | REL-1017
Number analyzed (Participants) | 186
mmHg | 0.0 (10.9)

9. Secondary Outcome: Change in Heart Rate From Baseline to Month 3
Description: Cardiac Safety of REL-1017 as measured by the Heart Rate (Supine/Semi-Supine) From Baseline to Month 3.
  A negative change from baseline indicates a reduction in Heart Rate.
Time Frame: 3 Month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | REL-1017
Number analyzed (Participants) | 505
beats/min | 0.8 (9.2)

10. Secondary Outcome: Change in Heart Rate From Baseline to Month 12
Description: Cardiac Safety of REL-1017 as measured by the Heart Rate (Supine/Semi-Supine) From Baseline to Month 12.
  A negative change from baseline indicates a reduction in Heart Rate.
Time Frame: 12 Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | REL-1017
Number analyzed (Participants) | 186
beats/min | -0.1 (9.6)

11. Secondary Outcome: Change in Weight From Baseline to Month 3
Description: Overall Safety of REL-1017 as measured by Weight From Baseline to Month 3.
  A negative change from baseline indicates a reduction in Weight.
Time Frame: 3 Month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | REL-1017
Number analyzed (Participants) | 545
kg | 0.32 (4.45)

12. Secondary Outcome: Change in Weight From Baseline to Month 12
Description: Overall Safety of REL-1017 as measured by Weight From Baseline to Month 12.
  A negative change from baseline indicates a reduction in Weight.
Time Frame: 12 Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | REL-1017
Number analyzed (Participants) | 197
kg | 0.33 (5.56)

13. Other Pre Specified Outcome: Change in the MADRS10 Total Score From Baseline to Month 3
Description: Therapeutic efficacy of REL-1017 in the Montgomery-Asberg Depression Rating Scale (MADRS10) A higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60 with scores above 34 indicating severe depression.
  A negative change from baseline indicates improvement.
Time Frame: 3 Month
Population: Full Analysis Set (FAS) at Month 3: All participants who received at least 1 dose of study drug and had at least one post-Baseline efficacy assessment, irrespective of any deviation from the protocol or premature discontinuation at Month 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REL-1017
Number analyzed (Participants) | 536
units on a scale | -20.1 (10.7)

14. Other Pre Specified Outcome: Change in the MADRS10 Total Score From Baseline to Month 12
Description: as for outcome 13
Time Frame: 12 Month
Population: Full Analysis Set (FAS) at Month 12: All participants who received at least 1 dose of study drug and had at least one post-Baseline efficacy assessment, irrespective of any deviation from the protocol or premature discontinuation at Month 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REL-1017
Number analyzed (Participants) | 199
units on a scale | -21.6 (10.4)

ADVERSE EVENTS:
Time Frame: A Treatment Emergent Adverse Event (TEAE) is defined as an Adverse Event (AE) that starts or worsens at any time after initiation of study drug collected up to 1 month post treatment (Day 395) as collected in the Safety Analysis Set.
Description: A TEAE is defined as an AE that starts or worsens at any time after initiation of study drug collected up to 1 month post treatment (Day 395) as collected in the Safety Analysis Set.
Arm/Group | REL-1017
All-Cause Mortality (participants affected / at risk) | 0/624
Serious Adverse Events (participants affected / at risk) | 8/624
Other Adverse Events (participants affected / at risk) | 142/624
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REL-1017 (N=624)
Coronary artery disease (Cardiac disorders) | 1 (1) — Not related to study drug.
Tachycardia (Cardiac disorders) | 1 (1) — Not related to study drug.
Alcohol abuse (Psychiatric disorders) | 1 (1) — Not related to study drug.
Anxiety (Psychiatric disorders) | 1 (1) — Not related to study drug.
Anaphylactic reaction (Immune system disorders) | 1 (1) — Not related to study drug.
Bacteraemia (Infections and infestations) | 1 (1) — Not related to study drug.
Pyelonephritis (Infections and infestations) | 1 (1) — Not related to study drug.
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) — Not related to study drug.
Hyperreflexia (Nervous system disorders) | 1 (1) — Not related to study drug.
Tremor (Nervous system disorders) | 1 (1) — Not related to study drug.
Sepsis (Infections and infestations) | 1 (1) — Not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REL-1017 (N=624)
COVID-19 (Infections and infestations) | 60 (62) — Not related to study drug.
Headache (Nervous system disorders) | 61 (77)
Upper respiratory tract infections (Infections and infestations) | 53 (67) — Not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT04855760/Prot_SAP_000.pdf